CLINICAL TRIAL: NCT00526669
Title: An Exploratory, Phase II Trial to Determine the Association of Lapatinib Induced Fluoropyrimidine Gene Changes With Efficacy Parameters of Lapatinib and Capecitabine in First Line Gastric Cancer
Brief Title: Study For Patients With Untreated Gastric Cancer Who Will Receive Capecitabine And Lapatinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPT109747
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Results first posted 2012-10-01 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-07

CONDITIONS: Neoplasms, Gastrointestinal Tract
Keywords: tumor biopsy; capecitabine; first line; Gastro Esophageal (GE) Junction Cancer; Gastric cancer; newly diagnosed; GE junction; lapatinib; metastatic or unresectable
MeSH Terms: conditions — Neoplasms; Stomach Neoplasms; Neoplasm Metastasis | interventions — Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lapatinib and Capecitabine — oral lapatinib (1250mg) administered as a monotherapy run-in followed by its combination with capecitabine

SUMMARY:
The study will determine if changes in expression of markers involved in the 5-FU pathways are associated with response to treatment with the combination of lapatinib and capecitabine independent of tumor erbB2 status.

ELIGIBILITY:
Inclusion Criteria:

* Has signed inform consent
* Untreated, newly diagnosed, advanced metastatic or unresectable gastric cancer, including the gastro-esophageal junction
* Tumor accessible to and patient consent for endoscopic biopsy at study start and after 7 days of single agent Lapatinib
* Measurable disease according to RECIST criteria
* Male or female > or = 18 years of age
* Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram
* must have adequate organ function as defined by baseline laboratory values

Exclusion Criteria:

* Gastric carcinoid, sarcomas, or squamous cell cancer
* Pregnant or lactating females
* Intractable nausea, vomiting, or gastro intestinal obstruction requiring decompression and drainage with a gastric tube or nasogastric suction.
* patients who require continuous enteral feeding
* Malabsorption syndrome or uncontrolled inflammatory GI disease (Crohn's or ulcerative colitis
* Known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-03; Primary Completion 2011-04 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (19):
- United States (8):
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Southgate, Michigan
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Dallas, Texas
- GSK Investigational Site, Montreal, Quebec, Canada
- GSK Investigational Site, Mexico City, Mexico
- Russia (4):
  - GSK Investigational Site, Astrakhan
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Ufa
- South Korea (3):
  - GSK Investigational Site, Hwasun
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Gyeonggi-do
- Taiwan (2):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Taipei

REFERENCES:
- [Derived] LaBonte MJ, Yang D, Zhang W, Wilson PM, Nagarwala YM, Koch KM, Briner C, Kaneko T, Rha SY, Gladkov O, Urba SG, Sakaeva D, Pishvaian MJ, Hsieh RK, Lee WP, Lenz HJ. A Phase II Biomarker-Embedded Study of Lapatinib plus Capecitabine as First-line Therapy in Patients with Advanced or Metastatic Gastric Cancer. Mol Cancer Ther. 2016 Sep;15(9):2251-8. doi: 10.1158/1535-7163.MCT-15-0908. Epub 2016 Jun 20. PMID 27325685

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 68 participants were enrolled in the study, as reflected by the enrollment number in the protocol record; however, one participant elected to not receive study treatment and was thus not included in the Intent-to-Treat Population.
Pre-assignment Details: After an initial tumor biopsy (biop.), participants (par.) received lapatinib monotherapy in a 7-day Run-in Period, followed by a second biop. After the second biop., par. received a 14-day course of capecitabine in combination with lapatinib, which continued in the absence of treatment-related toxicity, until disease progression or withdrawal.
Groups:
- Lapatinib: Lapatinib 250 milligram (mg) tablets administered at a dose of 1250 mg once daily (OD) for 7 days
- Lapatinib + Capecitabine: Lapatinib tablets were administered orally at a dose of 1250 mg OD and capecitabine tablets were administered orally at a dose of 1000 milligrams per meters squared (mg/m^2) twice daily (BID) for the first 14 days of each subsequent 21-day cycle. The capecitabine dose schedule was an intermittent regimen consisting of 2 weeks of treatment followed by 1 week of rest (drug-free period). Capecitabine and lapatinib were taken at two different times of the day.
Period: 7-Day Run-in Monotherapy Treatment Phase
Arm/Group | Lapatinib | Lapatinib + Capecitabine
Started | 67 | 0
Completed | 67 | 0
Not Completed | 0 | 0
Period: Combined Treatment Phase
Arm/Group | Lapatinib | Lapatinib + Capecitabine
Started | 0 | 67
Completed | 0 | 59
Not Completed | 0 | 8
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Sponsor Terminated Study | 0 | 2
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data were collected in members of the Intent-to-Treat Population, comprised of all participants who entered the study and received at least one dose of lapatinib.
  Years | 61.4 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline data were collected in members of the Intent-to-Treat Population, comprised of all participants who entered the study and received at least one dose of lapatinib.
  Participants
    Female | 17
    Male | 50
Race/Ethnicity, Customized [Number; unit: participants] — Baseline data were collected in members of the Intent-to-Treat Population, comprised of all participants who entered the study and received at least one dose of lapatinib.
  participants
    White - White/Caucasian/European Heritage | 34
    Asian - East Asian Heritage | 30
    American Indian or Alaskan Native | 2
    Asian - South East Asian Heritage | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Start of Run-in Period in Biomarker Expression Levels at Day 0
Description: Participants were analyzed for intratumoral expression levels of genes involved in the 5-fluorouracil (FU) pathway and lapatinib-targeted genes. Change in biomarker expression levels was calculated as the levels measured after the lapatinib Run-in Period (Baseline) of the study minus the levels measured at the start of monotherapy (Day -7). EGFR, epidermal growth factor receptor; HER, human epidermal growth factor receptor. Data are presented as ratios of the normalized gene expression of the target gene to that of beta actin.
Time Frame: evaluated at baseline and after 7 days of study treatment
Population: Intent-to-Treat (ITT) Population: all participants who entered the study and received at least one dose of lapatinib. Only those participants contributing viable samples were analyzed. Different participants contributed samples for different biomarkers.
Measure: Median (Full Range); unit: ratio
Arm/Group | Lapatinib
Number analyzed (Participants) | 67
ratio
  Thymidylate synthase (TS), n=34 | 0.38 [-2.33 to 7.25]
  Deoxypyridinoline (DPD), n=26 | 0.12 [-0.61 to 1.04]
  EGFR/HER1, n=32 | 0.15 [-1.88 to 41.89]
  HER2, n=28 | 0.01 [-0.29 to 1.61]
  HER3, n=33 | 0.87 [-36.31 to 8.18]
Statistical Analysis 1: Comparison: Lapatinib; Test type: Superiority or Other; p = 0.10, Wilcoxon signed rank test — Biomarker: TS
Statistical Analysis 2: Comparison: Lapatinib; Test type: Superiority or Other; p = 0.097, Wilcoxon signed rank test — Biomarker: DPD
Statistical Analysis 3: Comparison: Lapatinib; Test type: Superiority or Other; p = 0.10, Wilcoxon signed rank test — Biomarker: EGFR/HER1
Statistical Analysis 4: Comparison: Lapatinib; Test type: Superiority or Other; p = 0.26, Wilcoxon signed rank test — Biomarker: HER2
Statistical Analysis 5: Comparison: Lapatinib; Test type: Superiority or Other; p = 0.38, Wilcoxon signed rank test — Biomarker: HER3

2. Primary Outcome: Response Rate (Measured as the Percentage of Participants With Response [Complete Response or Partial Response])
Description: Response is defined as documented evidence of complete response (CR) or partial response (PR). The investigator evaluated response based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Complete response is defined as the disappearance of all target lesions (TLs) and non-TLs and the appearance of no new lesions (NLs). Partial response for TLs is defined as >= a 30% decrease in the sum of the longest diameter (LD) of TLs, taking as a reference the Baseline sum LD. For non-TLs it is defined as the persistence of 1 or more non-TL and no new TLs or non-TLs.
Time Frame: From Baseline (Day 0) until disease progression or death due to any cause evaluated every 6 or 12 weeks (up to approximately 85 weeks)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 67
percentage of participants | 17.9
Statistical Analysis 1: Comparison: Lapatinib + Capecitabine; Test type: Superiority or Other; percentage of participants = 17.9, 95% CI 2-sided [9.6 to 29.2] — The estimated value represents the percentage of participants with complete response or partial response

3. Primary Outcome: Percentage of Participants (Par.) With 5-month Progression-free Survival (PFS)
Description: 5-month (mo.) PFS was defined as the percentage of par. who were alive/progression free for 5 months from the time of initial treatment. PFS is defined as the time from the initial treatment until the first observation of disease progression (DP)/death due to any cause; the percentage of par. whose follow-up ended or was ongoing was reported. DP is defined as symptomatic progression or the appearance of >=1 NL and/or unequivocal progression of existing non-TLs, and a >=20% increase in the sum of the LD of TLs, taking as a reference the smallest sum LD recorded since treatment started.
Time Frame: From initial treatment up to 24 weeks (next available assessment after the 5-month assessment for progressive disease)
Population: ITT Population. PFS was censored for participants who did not have an event before data cut off. The last available assessment prior to the data cut off was used for censored participants.
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 67
percentage of participants | 29
Statistical Analysis 1: Comparison: Lapatinib + Capecitabine; Test type: Superiority or Other; percentage of participants = 29, 95% CI 2-sided [17.9 to 40.3] — The estimated value reflects the percentage of participants who achieved progression-free survival

4. Secondary Outcome: PFS
Description: PFS is defined as the time from the initial treatment until the first observation of disease progression or death due to any cause. The date of documented disease progression was defined as the earliest date of radiographic disease assessment progression or symptomatic progression, whichever came first. For participants who did not die/progress, survival was censored at the time of the last assessment (or contact).
Time Frame: From Baseline (Day 0) until disease progression or death due to any cause (up to approximately 85 weeks)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 67
weeks | 14.3 [12.6 to 18.7]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the initial treatment until death due to any cause. A death occurring during the study is defined as a death occurring during treatment or within 30 days of the last administration of study medication.
Time Frame: From Baseline (Day 0) until death due to any cause evaluated at approximately 12 months (up to approximately 100 weeks)
Population: ITT Population. OS was censored for participants who did not have an event before data cut off. The last available assessment prior to the data cut off was used for censored participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 67
weeks | 27.6 [21.7 to 39.4]

6. Secondary Outcome: Time to Progression (All Deaths Are Treated as Competing Risk)
Description: Time to progression is defined as the time from the initial treatment (first dose) until the first documented radiological symptomatic sign of disease progression. Time to progression data are presented as cumulative incidence estimate, which is defined as the time from the initial treatment until crude hazard probability of the occurrence of a particular event is reached to a particular point. All factors that hinder the observation of the event are defined as competing risks.
Time Frame: From Baseline (Day 0) until disease progression or death due to any cause (up to approximately 85 weeks)
Population: ITT Population. Time to progression was censored for participants who did not have an event before data cut off. The last available assessment prior to the data cut off was used for censored participants.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 67
weeks | 18.9 [7.7 to 56.7]

7. Secondary Outcome: Time to Progression (All Deaths Due to Non-PD Are Treated as Competing Risk)
Description: Time to progression is defined as the time from the initial treatment (first dose) until the first documented radiological symptomatic sign of disease progression. Time to progression data are presented as cumulative incidence estimate, which is defined as the time from the initial treatment until crude hazard probability of occurrence of a particular event is reached to a particular point. All factors that hinder the observation of the event are defined as competing risks.
Time Frame: From Baseline (Day 0) until disease progression or death due to any cause (up to approximately 85 weeks)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 67
weeks | 14.3 [7.4 to 24.9]

8. Secondary Outcome: Time to Response
Description: Time to response is defined as the time from the initial treatment until the first documented evidence of CR (disappearance of all TLs and non-TLs and the appearance of no new lesions) or PR (>= a 30% decrease in the sum of the longest diameter of TLs, taking as reference the Baseline sum longest diameter) (whichever status was recorded first). Time to response data are presented as cumulative incidence estimate, which is defined as the time from the initial treatment until crude hazard probability of the occurrence of a particular event is reached to a particular point.
Time Frame: Baseline (Day 0) until first documented evidence of response (up to approximately 60 weeks)
Population: ITT Population. Time to response was censored for participants who did not have an event before data cut off. The last available assessment prior to the data cut off was used for censored participants.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 67
weeks | NA [NA to NA] — Insufficient numbers of responses were observed; therefore, the median and the inter-quartile range cannot be estimated.

9. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the first documented evidence of tumor response (CR or PR) until the first documented sign of disease progression or death due to any cause, whichever came first.
Time Frame: From date of first documented evidence of response until the date of first documented sign of disease progression or death due to any cause (up to approximately 78 weeks)
Population: ITT Population. Duration of response was estimated for only the subset of participants who had response. Duration of response was censored for participants who did not have an event before data cut off. The last available assessment prior to the data cut off was used for censored participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 12
weeks | 18.4 [12.3 to 36.0]

10. Secondary Outcome: Number of Participants in the Indicated Categories for Best Overall Response (BOR)
Description: Best overall response was evaluated by the investigator based on RECIST criteria: CR; PR; Stable Disease (SD), defined as no sufficient shrinkage to qualify for PR, no sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum LD since the treatment started; PD, defined as at least a 20% increase in the sum of the LD of target lesions, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of >= 1 new lesions; Unknown, defined as participants who do not have CR, PR, SD, or PD.
Time Frame: From Baseline (Day 0) until disease progression or death due to any cause (up to approximately 85 weeks)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 67
participants
  CR | 0
  PR | 12
  SD | 31
  PD | 16
  Unknown | 8

11. Secondary Outcome: Number of Participants With Change From Baseline (Measured as Any Grade Increase [AGI], Increase to Grade 3 [ItoG3], and Increase to Grade 4 [ItoG4]) in Toxicity Grades for Albumin at the Indicated Time Points
Description: Toxicity was measured in grades (AE severity) per National Cancer Institute Common Toxicity Criteria for Adverse Event (NCI CTCAE) version (v) 3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For albumin (per blood samples): G 1 (<lower limit of normal [LLN] to 3 grams per deciliter [g/dL]), mild; G 2 (<3 to 2 g/dL), moderate; G 3 (<2 g/dL), severe; G 4 (value not available), life threatening/disabling; G 5 (death), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: Baseline (Day 0); Weeks 1, 2, 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, and 84; withdrawal (WD)/study conclusion (up to approximately 87 weeks); and worst-case on-therapy
Population: Safety Population: all participants who entered the study and received at least one dose of lapatinib. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 65
participants
  Week 1, AGI; n=54 | 10
  Week 2, AGI; n=57 | 9
  Week 3, AGI; n=61 | 10
  Week 6, AGI; n=47 | 4
  Week 9, AGI; n=41 | 2
  Week 12, AGI; n=31 | 4
  Week 15, AGI; n=22 | 3
  Week 18, AGI; n=17 | 1
  Week 21, AGI; n=14 | 1
  Week 24, AGI; n=11 | 1
  Week 30, AGI; n=9 | 0
  Week 36, AGI; n=5 | 0
  Week 42, AGI; n=4 | 0
  Week 48, AGI; n=3 | 0
  Week 54, AGI; n=3 | 0
  Week 60, AGI; n=2 | 1
  Week 66, AGI; n=1 | 0
  Week 72, AGI; n=1 | 0
  Week 78, AGI; n=1 | 0
  Week 84, AGI; n=1 | 0
  Withdrawal /study conclusion, AGI; n=50 | 11
  Worst-case on-therapy, AGI; n=65 | 29
  Week 1, ItoG3; n=54 | 0
  Week 2, ItoG3; n=57 | 0
  Week 3, ItoG3; n=61 | 0
  Week 6, ItoG3; n=47 | 0
  Week 9, ItoG3; n=41 | 0
  Week 12, ItoG3; n=31 | 0
  Week 15, ItoG3; n=22 | 0
  Week 18, ItoG3; n=17 | 0
  Week 21, ItoG3; n=14 | 0
  Week 24, ItoG3; n=11 | 0
  Week 30, ItoG3; n=9 | 0
  Week 36, ItoG3; n=5 | 0
  Week 42, ItoG3; n=4 | 0
  Week 48, ItoG3; n=3 | 0
  Week 54, ItoG3; n=3 | 0
  Week 60, ItoG3; n=2 | 0
  Week 66, ItoG3; n=1 | 0
  Week 72, ItoG3; n=1 | 0
  Week 78, ItoG3; n=1 | 0
  Week 84, ItoG3; n=1 | 0
  WD/study conclusion, ItoG3; n=50 | 0
  Worst-case on-therapy, ItoG3; n=65 | 0
  Week 1, ItoG4; n=54 | 0
  Week 2, ItoG4; n=57 | 0
  Week 3, ItoG4; n=61 | 0
  Week 6, ItoG4; n=47 | 0
  Week 9, ItoG4; n=41 | 0
  Week 12, ItoG4; n=31 | 0
  Week 15, ItoG4; n=22 | 0
  Week 18, ItoG4; n=17 | 0
  Week 21, ItoG4; n=14 | 0
  Week 24, ItoG4; n=11 | 0
  Week 30, ItoG4; n=9 | 0
  Week 36, ItoG4; n=5 | 0
  Week 42, ItoG4; n=4 | 0
  Week 48, ItoG4; n=3 | 0
  Week 54, ItoG4; n=3 | 0
  Week 60, ItoG4; n=2 | 0
  Week 66, ItoG4; n=1 | 0
  Week 72, ItoG4; n=1 | 0
  Week 78, ItoG4; n=1 | 0
  Week 84, ItoG4; n=1 | 0
  WD/study conclusion, ItoG4; n=50 | 0
  Worst-case on-therapy ItoG4; n=65 | 0

12. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4) in Toxicity Grades for Alkaline Phosphatase (ALP) at the Indicated Time Points
Description: Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For ALP: G 1 (upper limit of normal [ULN] to 2.5x ULN), mild; G 2 (>2.5 to 5.0x ULN), moderate; G 3 (>5.0 to 20.0x ULN), severe; G 4 (>20.0x ULN), life threatening/disabling; G 5 (value not available), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 65
participants
  Week 1, AGI; n=54 | 6
  Week 2, AGI; n=57 | 5
  Week 3, AGI; n=61 | 8
  Week 6, AGI; n=47 | 5
  Week 9, AGI; n=41 | 2
  Week 12, AGI; n=31 | 5
  Week 15, AGI; n=22 | 2
  Week 18, AGI; n=17 | 3
  Week 21, AGI; n=14 | 4
  Week 24, AGI; n=11 | 4
  Week 30, AGI; n=9 | 3
  Week 36, AGI; n=5 | 1
  Week 42, AGI; n=4 | 1
  Week 48, AGI; n=3 | 1
  Week 54, AGI; n=2 | 2
  Week 60, AGI; n=2 | 1
  Week 66, AGI; n=1 | 1
  Week 72, AGI; n=1 | 1
  Week 78, AGI; n=1 | 1
  Week 84, AGI; n=1 | 1
  WD/study conclusion, AGI; n=49 | 8
  Worst-case on-therapy, AGI; n=65 | 21
  Week 1, ItoG3; n=54 | 0
  Week 2, ItoG3; n=57 | 0
  Week 3, ItoG3; n=61 | 0
  Week 6, ItoG3; n=47 | 0
  Week 9, ItoG3; n=41 | 0
  Week 12, ItoG3; n=31 | 0
  Week 15, ItoG3; n=22 | 0
  Week 18, ItoG3; n=17 | 0
  Week 21, ItoG3; n=14 | 1
  Week 24, ItoG3; n=11 | 0
  Week 30, ItoG3; n=9 | 0
  Week 36, ItoG3; n=5 | 0
  Week 42, ItoG3; n=4 | 0
  Week 48, ItoG3; n=3 | 0
  Week 54, ItoG3; n=2 | 0
  Week 60, ItoG3; n=2 | 0
  Week 66, ItoG3; n=1 | 0
  Week 72, ItoG3; n=1 | 0
  Week 78, ItoG3; n=1 | 0
  Week 84, ItoG3; n=1 | 0
  WD/study conclusion, ItoG3; n=49 | 1
  Worst-case on-therapy, ItoG3; n=65 | 2
  Week 1, ItoG4; n=54 | 0
  Week 2, ItoG4; n=57 | 0
  Week 3, ItoG4; n=61 | 0
  Week 6, ItoG4; n=47 | 0
  Week 9, ItoG4; n=41 | 0
  Week 12, ItoG4; n=31 | 0
  Week 15, ItoG4; n=22 | 0
  Week 18, ItoG4; n=17 | 0
  Week 21, ItoG4; n=14 | 0
  Week 24, ItoG4; n=11 | 0
  Week 30, ItoG4; n=9 | 0
  Week 36, ItoG4; n=5 | 0
  Week 42, ItoG4; n=4 | 0
  Week 48, ItoG4; n=3 | 0
  Week 54, ItoG4; n=2 | 0
  Week 60, ItoG4; n=2 | 0
  Week 66, ItoG4; n=1 | 0
  Week 72, ItoG4; n=1 | 0
  Week 78, ItoG4; n=1 | 0
  Week 84, ItoG4; n=1 | 0
  WD/study conclusion, ItoG4; n=49 | 0
  Worst-case on-therapy, ItoG4; n=65 | 0

13. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4) in Toxicity Grades for Aspartate Aminotransferase (AST) at the Indicated Time Points
Description: Blood samples were collected for the evaluation of AST. Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For AST: G 1 (>ULN to 2.5x ULN), mild; G 2 (>2.5 to 5.0x ULN), moderate; G 3 (>5.0 to 20.0x ULN), severe; G 4 (>20.0x ULN), life threatening/disabling; G 5 (value not available), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 65
participants
  Week 1, AGI; n=54 | 1
  Week 2, AGI; n=57 | 3
  Week 3, AGI; n=61 | 3
  Week 6, AGI; n=47 | 6
  Week 9, AGI; n=41 | 3
  Week 12, AGI; n=31 | 2
  Week 15, AGI; n=22 | 4
  Week 18, AGI; n=17 | 1
  Week 21, AGI; n=14 | 1
  Week 24, AGI; n=11 | 0
  Week 30, AGI; n=9 | 2
  Week 36, AGI; n=5 | 0
  Week 42, AGI; n=4 | 0
  Week 48, AGI; n=3 | 0
  Week 54, AGI; n=3 | 0
  Week 60, AGI; n=2 | 0
  Week 66, AGI; n=1 | 0
  Week 72, AGI; n=1 | 0
  Week 78, AGI; n=1 | 0
  Week 84, AGI; n=1 | 1
  WD/study conclusion, AGI; n=50 | 7
  Worst-case on-therapy, AGI; n=65 | 16
  Week 1, ItoG3; n=54 | 0
  Week 2, ItoG3; n=57 | 0
  Week 3, ItoG3; n=61 | 0
  Week 6, ItoG3; n=47 | 0
  Week 9, ItoG3; n=41 | 0
  Week 12, ItoG3; n=31 | 0
  Week 15, ItoG3; n=22 | 0
  Week 18, ItoG3; n=17 | 0
  Week 21, ItoG3; n=14 | 0
  Week 24, ItoG3; n=11 | 0
  Week 30, ItoG3; n=9 | 0
  Week 36, ItoG3; n=5 | 0
  Week 42, ItoG3; n=4 | 0
  Week 48, ItoG3; n=3 | 0
  Week 54, ItoG3; n=3 | 0
  Week 60, ItoG3I; n=2 | 0
  Week 66, ItoG3; n=1 | 0
  Week 72, ItoG3; n=1 | 0
  Week 78, ItoG3; n=1 | 0
  Week 84, ItoG3; n=1 | 0
  WD/study conclusion, ItoG3; n=50 | 1
  Worst-case on-therapy, ItoG3; n=65 | 1
  Week 1, ItoG4; n=54 | 0
  Week 2, ItoG4; n=57 | 0
  Week 3, ItoG4; n=61 | 0
  Week 6, ItoG4; n=47 | 0
  Week 9, ItoG4; n=41 | 0
  Week 12, ItoG4; n=31 | 0
  Week 15, ItoG4; n=22 | 0
  Week 18, ItoG4; n=17 | 0
  Week 21, ItoG4; n=14 | 0
  Week 24, ItoG4; n=11 | 0
  Week 30, ItoG4; n=9 | 0
  Week 36, ItoG4; n=5 | 0
  Week 42, ItoG4; n=4 | 0
  Week 48, ItoG4; n=3 | 0
  Week 54, ItoG4; n=3 | 0
  Week 60, ItoG4; n=2 | 0
  Week 66, ItoG4; n=1 | 0
  Week 72, ItoG4; n=1 | 0
  Week 78, ItoG4; n=1 | 0
  Week 84, ItoG4; n=1 | 0
  WD/study conclusion, ItoG4; n=50 | 0
  Worst-case on-therapy, ItoG4; n=65 | 0

14. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4 ) in Toxicity Grades for Alanine Aminotransferase (ALT) at the Indicated Time Points
Description: Blood samples were collected for the evaluation of ALT. Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For ALT: G 1 (>ULN to 2.5x ULN), mild; G 2 (>2.5 to 5.0x ULN), moderate; G 3 (>5.0 to 20.0x ULN), severe; G 4 (>20.0x ULN), life threatening/disabling; G 5 (value not available), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 65
participants
  Week 1, AGI; n=54 | 1
  Week 2, AGI; n=57 | 0
  Week 3, AGI; n=61 | 2
  Week 6, AGI; n=47 | 3
  Week 9, AGI; n=41 | 2
  Week 12, AGI; n=31 | 2
  Week 15, AGI; n=22 | 2
  Week 18, AGI; n=17 | 0
  Week 21, AGI; n=14 | 0
  Week 24, AGI; n=11 | 0
  Week 30, AGI; n=9 | 0
  Week 36, AGI; n=5 | 0
  Week 42, AGI; n=4 | 0
  Week 48, AGI; n=3 | 0
  Week 54, AGI; n=3 | 0
  Week 60, AGI; n=2 | 0
  Week 66, AGI; n=1 | 0
  Week 72, AGI; n=1 | 0
  Week 78, AGI; n=1 | 0
  Week 84, AGI; n=1 | 0
  WD/study conclusion, AGI; n=50 | 0
  Worst-case on-therapy, AGI; n=65 | 10
  Week 1, ItoG3; n=54 | 0
  Week 2, ItoG3; n=57 | 0
  Week 3, ItoG3; n=61 | 0
  Week 6, ItoG3; n=47 | 0
  Week 9, ItoG3; n=41 | 0
  Week 12, ItoG3; n=31 | 0
  Week 15, ItoG3; n=22 | 0
  Week 18, ItoG3; n=17 | 0
  Week 21, ItoG3; n=14 | 0
  Week 24, ItoG3; n=11 | 0
  Week 30, ItoG3; n=9 | 0
  Week 36, ItoG3; n=5 | 0
  Week 42, ItoG3; n=4 | 0
  Week 48, ItoG3; n=3 | 0
  Week 54, ItoG3; n=3 | 0
  Week 60, ItoG3I; n=2 | 0
  Week 66, ItoG3; n=1 | 0
  Week 72, ItoG3; n=1 | 0
  Week 78, ItoG3; n=1 | 0
  Week 84, ItoG3; n=1 | 0
  WD/study conclusion, ItoG3; n=50 | 1
  Worst-case on-therapy, ItoG3; n=65 | 1
  Week 1, ItoG4; n=54 | 0
  Week 2, ItoG4; n=57 | 0
  Week 3, ItoG4; n=61 | 0
  Week 6, ItoG4; n=47 | 0
  Week 9, ItoG4; n=41 | 0
  Week 12, ItoG4; n=31 | 0
  Week 15, ItoG4; n=22 | 0
  Week 18, ItoG4; n=17 | 0
  Week 21, ItoG4; n=14 | 0
  Week 24, ItoG4; n=11 | 0
  Week 30, ItoG4; n=9 | 0
  Week 36, ItoG4; n=5 | 0
  Week 42, ItoG4; n=4 | 0
  Week 48, ItoG4; n=3 | 0
  Week 54, ItoG4; n=3 | 0
  Week 60, ItoG4; n=2 | 0
  Week 66, ItoG4; n=1 | 0
  Week 72, ItoG4; n=1 | 0
  Week 78, ItoG4; n=1 | 0
  Week 84, ItoG4; n=1 | 0
  WD/study conclusion, ItoG4; n=50 | 0
  Worst-case on-therapy, ItoG4; n=65 | 0

15. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4) in Toxicity Grades for Total Bilirubin at the Indicated Time Points
Description: Blood samples were collected for the evaluation of total bilirubin. Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For total bilirubin: G 1 (>ULN to 1.5x ULN), mild; G 2 (>1.5 to 3.0x ULN), moderate; G 3 (>3.0 to 10.0x ULN), severe; G 4 (>10.0x ULN), life threatening/disabling; G 5 (value not available), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 65
participants
  Week 1, AGI; n=54 | 0
  Week 2, AGI; n=57 | 2
  Week 3, AGI; n=61 | 1
  Week 6, AGI; n=47 | 2
  Week 9, AGI; n=41 | 8
  Week 12, AGI; n=31 | 3
  Week 15, AGI; n=22 | 3
  Week 18, AGI; n=17 | 2
  Week 21, AGI; n=14 | 3
  Week 24, AGI; n=11 | 3
  Week 30, AGI; n=9 | 4
  Week 36, AGI; n=5 | 1
  Week 42, AGI; n=4 | 1
  Week 48, AGI; n=3 | 1
  Week 54, AGI; n=3 | 0
  Week 60, AGI; n=2 | 0
  Week 66, AGI; n=1 | 0
  Week 72, AGI; n=1 | 1
  Week 78, AGI; n=1 | 0
  Week 84, AGI; n=1 | 1
  WD/study conclusion, AGI; n=50 | 4
  Worst-case on-therapy, AGI; n=65 | 13
  Week 1, ItoG3; n=54 | 0
  Week 2, ItoG3; n=57 | 0
  Week 3, ItoG3; n=61 | 0
  Week 6, ItoG3; n=47 | 0
  Week 9, ItoG3; n=41 | 0
  Week 12, ItoG3; n=31 | 0
  Week 15, ItoG3; n=22 | 0
  Week 18, ItoG3; n=17 | 0
  Week 21, ItoG3; n=14 | 0
  Week 24, ItoG3; n=11 | 0
  Week 30, ItoG3; n=9 | 0
  Week 36, ItoG3; n=5 | 0
  Week 42, ItoG3; n=4 | 0
  Week 48, ItoG3; n=3 | 0
  Week 54, ItoG3; n=3 | 0
  Week 60, ItoG3I; n=2 | 0
  Week 66, ItoG3; n=1 | 0
  Week 72, ItoG3; n=1 | 0
  Week 78, ItoG3; n=1 | 0
  Week 84, ItoG3; n=1 | 0
  WD/study conclusion, ItoG3; n=50 | 1
  Worst-case on-therapy, ItoG3; n=65 | 1
  Week 1, ItoG4; n=54 | 0
  Week 2, ItoG4; n=57 | 0
  Week 3, ItoG4; n=61 | 0
  Week 6, ItoG4; n=47 | 0
  Week 9, ItoG4; n=41 | 0
  Week 12, ItoG4; n=31 | 0
  Week 15, ItoG4; n=22 | 0
  Week 18, ItoG4; n=17 | 0
  Week 21, ItoG4; n=14 | 0
  Week 24, ItoG4; n=11 | 0
  Week 30, ItoG4; n=9 | 0
  Week 36, ItoG4; n=5 | 0
  Week 42, ItoG4; n=4 | 0
  Week 48, ItoG4; n=3 | 0
  Week 54, ItoG4; n=3 | 0
  Week 60, ItoG4; n=2 | 0
  Week 66, ItoG4; n=1 | 0
  Week 72, ItoG4; n=1 | 0
  Week 78, ItoG4; n=1 | 0
  Week 84, ItoG4; n=1 | 0
  WD/study conclusion, ItoG4; n=50 | 0
  Worst-case on-therapy, ItoG4; n=65 | 0

16. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4) in Toxicity Grades for Calcium at the Indicated Time Points
Description: Blood samples were collected for calcium evaluation. Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For calcium (low and high, respectively): G 1 (<LLN to 8.0 mg/dL; >ULN to 11.5x ULN), mild; G 2 (<8.0 to 7.0 mg/dL; >11.5 to 12.5 ULN), moderate; G 3 (<7.0 to 6.0 mg/dL; >12.5 to 13.5 mg/dL), severe; G 4 (<6 mg/dL; >13.5 mg/dL), life threatening/disabling; G 5 (death), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 65
participants
  Week 1, AGI; n=55 | 7
  Week 2, AGI; n=56 | 4
  Week 3, AGI; n=60 | 5
  Week 6, AGI; n=47 | 3
  Week 9, AGI; n=41 | 3
  Week 12, AGI; n=31 | 2
  Week 15, AGI; n=22 | 1
  Week 18, AGI; n=17 | 2
  Week 21, AGI; n=14 | 0
  Week 24, AGI; n=11 | 1
  Week 30, AGI; n=9 | 1
  Week 36, AGI; n=5 | 0
  Week 42, AGI; n=4 | 1
  Week 48, AGI; n=3 | 0
  Week 54, AGI; n=2 | 1
  Week 60, AGI; n=2 | 2
  Week 66, AGI; n=1 | 0
  Week 72, AGI; n=1 | 0
  Week 78, AGI; n=1 | 0
  Week 84, AGI; n=1 | 1
  WD/study conclusion, AGI; n=49 | 12
  Worst-case on-therapy, AGI; n=65 | 23
  Week 1, ItoG3; n=55 | 0
  Week 2, ItoG3; n=56 | 0
  Week 3, ItoG3; n=60 | 0
  Week 6, ItoG3; n=47 | 0
  Week 9, ItoG3; n=41 | 0
  Week 12, ItoG3; n=31 | 0
  Week 15, ItoG3; n=22 | 0
  Week 18, ItoG3; n=17 | 0
  Week 21, ItoG3; n=14 | 0
  Week 24, ItoG3; n=11 | 0
  Week 30, ItoG3; n=9 | 0
  Week 36, ItoG3; n=5 | 0
  Week 42, ItoG3; n=4 | 0
  Week 48, ItoG3; n=3 | 0
  Week 54, ItoG3; n=2 | 0
  Week 60, ItoG3; n=2 | 0
  Week 66, ItoG3; n=1 | 0
  Week 72, ItoG3; n=1 | 0
  Week 78, ItoG3; n=1 | 0
  Week 84, ItoG3; n=1 | 0
  WD/study conclusion, ItoG3; n=49 | 0
  Worst-case on-therapy, ItoG3; n=65 | 0
  Week 1, ItoG4; n=55 | 0
  Week 2, ItoG4; n=56 | 0
  Week 3, ItoG4; n=60 | 0
  Week 6, ItoG4; n=47 | 0
  Week 9, ItoG4; n=41 | 0
  Week 12, ItoG4; n=31 | 0
  Week 15, ItoG4; n=22 | 0
  Week 18, ItoG4; n=17 | 0
  Week 21, ItoG4; n=14 | 0
  Week 24, ItoG4; n=11 | 0
  Week 30, ItoG4; n=9 | 0
  Week 36, ItoG4; n=5 | 0
  Week 42, ItoG4; n=4 | 0
  Week 48, ItoG4; n=3 | 0
  Week 54, ItoG4; n=2 | 0
  Week 60, ItoG4; n=2 | 0
  Week 66, ItoG4; n=1 | 0
  Week 72, ItoG4; n=1 | 0
  Week 78, ItoG4; n=1 | 0
  Week 84, ItoG4; n=1 | 0
  WD/study conclusion, ItoG4; n=49 | 0
  Worst-case on-therapy, ItoG4; n=65 | 0

17. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4) in Toxicity Grades for Creatinine at the Indicated Time Points
Description: Blood samples were collected for the evaluation of creatinine. Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For creatinine: G 1 (>ULN to 1.5x ULN), mild; G 2 (>1.5 to 3.0x ULN), moderate; G 3 (>3.0 to 6.0x ULN), severe; G 4 (>6.0x ULN), life threatening/disabling; G 5 (death), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 65
participants
  Week 1, AGI; n=54 | 2
  Week 2, AGI; n=56 | 1
  Week 3, AGI; n=61 | 1
  Week 6, AGI; n=47 | 1
  Week 9, AGI; n=40 | 0
  Week 12, AGI; n=31 | 1
  Week 15, AGI; n=22 | 0
  Week 18, AGI; n=17 | 2
  Week 21, AGI; n=14 | 0
  Week 24, AGI; n=11 | 0
  Week 30, AGI; n=9 | 0
  Week 36, AGI; n=5 | 0
  Week 42, AGI; n=4 | 1
  Week 48, AGI; n=3 | 0
  Week 54, AGI; n=3 | 0
  Week 60, AGI; n=2 | 0
  Week 66, AGI; n=1 | 0
  Week 72, AGI; n=1 | 0
  Week 78, AGI; n=1 | 0
  Week 84 AGI; n=1 | 0
  WD/study conclusion, AGI; n=50 | 3
  Worst-case on-therapy, AGI; n=65 | 6
  Week 1, ItoG3; n=54 | 0
  Week 2, ItoG3; n=56 | 0
  Week 3, ItoG3; n=61 | 0
  Week 6, ItoG3; n=47 | 0
  Week 9, ItoG3; n=40 | 0
  Week 12, ItoG3; n=31 | 0
  Week 15, ItoG3; n=22 | 0
  Week 18, ItoG3; n=17 | 0
  Week 21, ItoG3; n=14 | 0
  Week 24, ItoG3; n=11 | 0
  Week 30, ItoG3; n=9 | 0
  Week 36, ItoG3; n=5 | 0
  Week 42, ItoG3; n=4 | 0
  Week 48, ItoG3; n=3 | 0
  Week 54, ItoG3; n=3 | 0
  Week 60, ItoG3; n=2 | 0
  Week 66, ItoG3; n=1 | 0
  Week 72, ItoG3; n=1 | 0
  Week 78, ItoG3; n=1 | 0
  Week 84, ItoG3; n=1 | 0
  WD/study conclusion, ItoG3; n=50 | 0
  Worst-case on-therapy, ItoG3; n=65 | 0
  Week 1, ItoG4; n=54 | 0
  Week 2, ItoG4; n=56 | 0
  Week 3, ItoG4; n=61 | 0
  Week 6, ItoG4; n=47 | 0
  Week 9, ItoG4; n=40 | 0
  Week 12, ItoG4; n=31 | 0
  Week 15, ItoG4; n=22 | 0
  Week 18, ItoG4; n=17 | 0
  Week 21, ItoG4; n=14 | 0
  Week 24, ItoG4; n=11 | 0
  Week 30, ItoG4; n=9 | 0
  Week 36, ItoG4; n=5 | 0
  Week 42, ItoG4; n=4 | 0
  Week 48, ItoG4; n=3 | 0
  Week 54, ItoG4; n=3 | 0
  Week 60, ItoG4; n=2 | 0
  Week 66, ItoG4; n=1 | 0
  Week 72, ItoG4; n=1 | 0
  Week 78, ItoG4; n=1 | 0
  Week 84, ItoG4; n=1 | 0
  WD/study conclusion, ItoG4; n=50 | 0
  Worst-case on-therapy, ItoG4; n=65 | 0

18. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4) in Toxicity Grades for Glucose at the Indicated Time Points
Description: Blood samples were collected for the evaluation of glucose. Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For glucose (high and low, respectively): G 1 (>ULN to 160 mg/dL; <LLN to 55 mg/dL), mild; G 2 (>160 to 250 mg/dL; <55 to 40 mg/dL), moderate; G 3 (>250 to 500 mg/dL; <40 to 30 mg/dL), severe; G 4 (>500 mg/dL; <30 mg/dL), life threatening/disabling; G 5 (death), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 65
participants
  Week 1, AGI; n=54 | 13
  Week 2, AGI; n=57 | 10
  Week 3, AGI; n=61 | 10
  Week 6, AGI; n=47 | 7
  Week 9, AGI; n=40 | 6
  Week 12, AGI; n=31 | 4
  Week 15, AGI; n=22 | 3
  Week 18, AGI; n=17 | 1
  Week 21, AGI; n=14 | 1
  Week 24, AGI; n=11 | 2
  Week 30, AGI; n=9 | 0
  Week 36, AGI; n=5 | 1
  Week 42, AGI; n=4 | 0
  Week 48, AGI; n=3 | 0
  Week 54, AGI; n=3 | 1
  Week 60, AGI; n=2 | 0
  Week 66, AGI; n=1 | 0
  Week 72, AGI; n=1 | 0
  Week 78, AGI; n=1 | 0
  Week 84, AGI; n=1 | 0
  WD/study conclusion, AGI; n=49 | 15
  Worst-case on-therapy, AGI; n=65 | 32
  Week 1, ItoG3; n=54 | 0
  Week 2, ItoG3; n=57 | 0
  Week 3, ItoG3; n=61 | 0
  Week 6, ItoG3; n=47 | 0
  Week 9, ItoG3; n=40 | 0
  Week 12, ItoG3; n=31 | 0
  Week 15, ItoG3; n=22 | 0
  Week 18, ItoG3; n=17 | 0
  Week 21, ItoG3; n=14 | 0
  Week 24, ItoG3; n=11 | 0
  Week 30, ItoG3; n=9 | 0
  Week 36, ItoG3; n=5 | 0
  Week 42, ItoG3; n=4 | 0
  Week 48, ItoG3; n=3 | 0
  Week 54, ItoG3; n=3 | 0
  Week 60, ItoG3; n=2 | 0
  Week 66, ItoG3; n=1 | 0
  Week 72, ItoG3; n=1 | 0
  Week 78, ItoG3; n=1 | 0
  Week 84, ItoG3; n=1 | 0
  WD/study conclusion, ItoG3; n=49 | 1
  Worst-case on-therapy, ItoG3; n=65 | 1
  Week 1, ItoG4; n=54 | 0
  Week 2, ItoG4; n=57 | 0
  Week 3, ItoG4; n=61 | 0
  Week 6, ItoG4; n=47 | 0
  Week 9, ItoG4; n=40 | 0
  Week 12, ItoG4; n=31 | 0
  Week 15, ItoG4; n=22 | 0
  Week 18, ItoG4; n=17 | 0
  Week 21, ItoG4; n=14 | 0
  Week 24, ItoG4; n=11 | 0
  Week 30, ItoG4; n=9 | 0
  Week 36, ItoG4; n=5 | 0
  Week 42, ItoG4; n=4 | 0
  Week 48, ItoG4; n=3 | 0
  Week 54, ItoG4; n=3 | 0
  Week 60, ItoG4; n=2 | 0
  Week 66, ItoG4; n=1 | 0
  Week 72, ItoG4; n=1 | 0
  Week 78, ItoG4; n=1 | 0
  Week 84, ItoG4; n=1 | 0
  WD/study conclusion, ItoG4; n=49 | 0
  Worst-case on-therapy, ItoG4; n=65 | 0

19. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4) in Toxicity Grades for Potassium at the Indicated Time Points
Description: Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For potassium (high and low [per blood samples], respectively): G 1 (>ULN to 5.5 millimoles per liter [mmol/L]; <LLN to 3.0 mmol/L), mild; G 2 (>5.5 to 6.0 mmol/L; value not available), moderate; G 3 (>6.0 to 7.0 mmol/L; <3.0 to 2.5 mmol/L), severe; G 4 (>7.0 mmol/L; <2.5 mmol/L), life threatening/disabling; G 5 (death), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 65
participants
  Week 1, AGI; n=54 | 9
  Week 2, AGI; n=54 | 3
  Week 3, AGI; n=59 | 5
  Week 6, AGI; n=46 | 3
  Week 9, AGI; n=41 | 4
  Week 12, AGI; n=31 | 4
  Week 15, AGI; n=22 | 1
  Week 18, AGI; n=17 | 2
  Week 21, AGI; n=13 | 1
  Week 24, AGI; n=11 | 0
  Week 30, AGI; n=9 | 2
  Week 36, AGI; n=5 | 0
  Week 42, AGI; n=4 | 0
  Week 48, AGI; n=3 | 0
  Week 54, AGI; n=3 | 0
  Week 60, AGI; n=2 | 0
  Week 66, AGI; n=1 | 0
  Week 72, AGI; n=1 | 0
  Week 78, AGI; n=1 | 0
  Week 84, AGI; n=1 | 0
  WD/study conclusion, AGI; n=48 | 7
  Worst-case on-therapy, AGI; n=65 | 25
  Week 1, ItoG3; n=54 | 1
  Week 2, ItoG3; n=54 | 0
  Week 3, ItoG3; n=59 | 1
  Week 6, ItoG3; n=46 | 0
  Week 9, ItoG3; n=41 | 0
  Week 12, ItoG3; n=31 | 0
  Week 15, ItoG3; n=22 | 0
  Week 18, ItoG3; n=17 | 0
  Week 21, ItoG3; n=13 | 0
  Week 24, ItoG3; n=11 | 0
  Week 30, ItoG3; n=9 | 0
  Week 36, ItoG3; n=5 | 0
  Week 42, ItoG3; n=4 | 0
  Week 48, ItoG3; n=3 | 0
  Week 54, ItoG3; n=3 | 0
  Week 60, ItoG3; n=2 | 0
  Week 66, ItoG3; n=1 | 0
  Week 72, ItoG3; n=1 | 0
  Week 78, ItoG3; n=1 | 0
  Week 84, ItoG3; n=1 | 0
  WD/study conclusion, ItoG3; n=48 | 2
  Worst-case on-therapy, ItoG3; n=65 | 5
  Week 1, ItoG4; n=54 | 0
  Week 2, ItoG4; n=54 | 0
  Week 3, ItoG4; n=59 | 0
  Week 6, ItoG4; n=46 | 0
  Week 9, ItoG4; n=41 | 1
  Week 12, ItoG4; n=31 | 0
  Week 15, ItoG4; n=22 | 0
  Week 18, ItoG4; n=17 | 0
  Week 21, ItoG4; n=13 | 0
  Week 24, ItoG4; n=11 | 0
  Week 30, ItoG4; n=9 | 0
  Week 36, ItoG4; n=5 | 0
  Week 42, ItoG4; n=4 | 0
  Week 48, ItoG4; n=3 | 0
  Week 54, ItoG4; n=3 | 0
  Week 60, ItoG4; n=2 | 0
  Week 66, ItoG4; n=1 | 0
  Week 72, ItoG4; n=1 | 0
  Week 78, ItoG4; n=1 | 0
  Week 84, ItoG4; n=1 | 0
  WD/study conclusion, ItoG4; n=48 | 0
  Worst-case on-therapy, ItoG4; n=65 | 1

20. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4) in Toxicity Grades for Magnesium at the Indicated Time Points
Description: Blood samples were collected for magnesium evaluation. Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For magnesium (high and low, respectively): G 1 (>ULN to 3.0 mg/dL; <LLN to 1.2 mg/dL), mild; G 2 (value not available; <1.2 to 0.9 mg/dL), moderate; G 3 (>3.0 to 8.0 mg/dL; <0.9 to 0.7 mg/dL), severe; G 4 (>8.0 mg/dL; <0.7 mg/dL), life threatening/disabling; G 5 (death), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 59
participants
  Week 1, AGI; n=33 | 1
  Week 2, AGI; n=33 | 6
  Week 3, AGI; n=44 | 3
  Week 6, AGI; n=37 | 4
  Week 9, AGI; n=36 | 1
  Week 12, AGI; n=27 | 0
  Week 15, AGI; n=18 | 1
  Week 18, AGI; n=16 | 1
  Week 21, AGI; n=11 | 0
  Week 24, AGI; n=9 | 0
  Week 30, AGI; n=9 | 0
  Week 36, AGI; n=5 | 0
  Week 42, AGI; n=4 | 0
  Week 48, AGI; n=3 | 0
  Week 54, AGI; n=2 | 0
  Week 60, AGI; n=2 | 0
  Week 66, AGI; n=1 | 0
  Week 72, AGI; n=1 | 0
  Week 78, AGI; n=1 | 0
  Week 84, AGI; n=1 | 0
  WD/study conclusion, AGI; n=35 | 6
  Worst-case on-therapy, AGI; n=59 | 17
  Week 1, ItoG3; n=33 | 0
  Week 2, ItoG3; n=33 | 0
  Week 3, ItoG3; n=44 | 0
  Week 6, ItoG3; n=37 | 1
  Week 9, ItoG3; n=36 | 0
  Week 12, ItoG3; n=27 | 0
  Week 15, ItoG3; n=18 | 0
  Week 18, ItoG3; n=16 | 0
  Week 21, ItoG3; n=11 | 0
  Week 24, ItoG3; n=9 | 0
  Week 30, ItoG3; n=9 | 0
  Week 36, ItoG3; n=5 | 0
  Week 42, ItoG3; n=4 | 0
  Week 48, ItoG3; n=3 | 0
  Week 54, ItoG3; n=2 | 0
  Week 60, ItoG3; n=2 | 0
  Week 66, ItoG3; n=1 | 0
  Week 72, ItoG3; n=1 | 0
  Week 78, ItoG3; n=1 | 0
  Week 84, ItoG3; n=1 | 0
  WD/study conclusion, ItoG3; n=35 | 1
  Worst-case on-therapy, ItoG3; n=59 | 2
  Week 1, ItoG4; n=33 | 0
  Week 2, ItoG4; n=33 | 0
  Week 3, ItoG4; n=44 | 0
  Week 6, ItoG4; n=37 | 0
  Week 9, ItoG4; n=36 | 0
  Week 12, ItoG4; n=27 | 0
  Week 15, ItoG4; n=18 | 0
  Week 18, ItoG4; n=16 | 0
  Week 21, ItoG4; n=11 | 0
  Week 24, ItoG4; n=9 | 0
  Week 30, ItoG4; n=9 | 0
  Week 36, ItoG4; n=5 | 0
  Week 42, ItoG4; n=4 | 0
  Week 48, ItoG4; n=3 | 0
  Week 54, ItoG4; n=2 | 0
  Week 60, ItoG4; n=2 | 0
  Week 66, ItoG4; n=1 | 0
  Week 72, ItoG4; n=1 | 0
  Week 78, ItoG4; n=1 | 0
  Week 84, ItoG4; n=1 | 0
  WD/study conclusion, ItoG4; n=35 | 0
  Worst-case on-therapy, ItoG4; n=59 | 0

21. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4) in Toxicity Grades for Sodium at the Indicated Time Points
Description: Blood samples were collected for sodium evaluation. Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of each AE severity. For sodium (high and low, respectively): G 1 (>ULN to 150 mmol/L; <LLN to 130 mmol/L), mild; G 2 (>150 to 155 mmol/L; value not available), moderate; G 3 (>155 to 160 mmol/L; <130 to 120 mmol/L), severe; G 4 (>160 mmol/L; <120 mmol/L), life threatening/disabling; G 5 (death), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 65
participants
  Week 1, AGI; n=54 | 9
  Week 2, AGI; n=53 | 7
  Week 3, AGI; n=59 | 5
  Week 6, AGI; n=47 | 7
  Week 9, AGI; n=41 | 4
  Week 12, AGI; n=31 | 1
  Week 15, AGI; n=22 | 3
  Week 18, AGI; n=17 | 1
  Week 21, AGI; n=13 | 0
  Week 24, AGI; n=11 | 1
  Week 30, AGI; n=9 | 2
  Week 36, AGI; n=5 | 0
  Week 42, AGI; n=4 | 0
  Week 48, AGI; n=3 | 0
  Week 54, AGI; n=3 | 0
  Week 60, AGI; n=2 | 0
  Week 66, AGI; n=1 | 0
  Week 72, AGI; n=1 | 0
  Week 78, AGI; n=1 | 0
  Week 84, AGI; n=1 | 0
  WD/study conclusion, AGI; n=48 | 10
  Worst-case on-therapy, AGI; n=65 | 28
  Week 1, ItoG3; n=54 | 0
  Week 2, ItoG3; n=53 | 1
  Week 3, ItoG3; n=59 | 0
  Week 6, ItoG3; n=47 | 0
  Week 9, ItoG3; n=41 | 1
  Week 12, ItoG3; n=31 | 0
  Week 15, ItoG3; n=22 | 0
  Week 18, ItoG3; n=17 | 0
  Week 21, ItoG3; n=13 | 0
  Week 24, ItoG3; n=11 | 0
  Week 30, ItoG3; n=9 | 1
  Week 36, ItoG3; n=5 | 0
  Week 42, ItoG3; n=4 | 0
  Week 48, ItoG3; n=3 | 0
  Week 54, ItoG3; n=3 | 0
  Week 60, ItoG3; n=2 | 0
  Week 66, ItoG3; n=1 | 0
  Week 72, ItoG3; n=1 | 0
  Week 78, ItoG3; n=1 | 0
  Week 84, ItoG3; n=1 | 0
  WD/study conclusion, ItoG3; n=48 | 2
  Worst-case on-therapy, ItoG3; n=65 | 4
  Week 1, ItoG4; n=54 | 1
  Week 2, ItoG4; n=53 | 0
  Week 3, ItoG4; n=59 | 0
  Week 6, ItoG4; n=47 | 0
  Week 9, ItoG4; n=41 | 0
  Week 12, ItoG4; n=31 | 0
  Week 15, ItoG4; n=22 | 0
  Week 18, ItoG4; n=17 | 0
  Week 21, ItoG4; n=13 | 0
  Week 24, ItoG4; n=11 | 0
  Week 30, ItoG4; n=9 | 0
  Week 36, ItoG4; n=5 | 0
  Week 42, ItoG4; n=4 | 0
  Week 48, ItoG4; n=3 | 0
  Week 54, ItoG4; n=3 | 0
  Week 60, ItoG4; n=2 | 0
  Week 66, ItoG4; n=1 | 0
  Week 72, ItoG4; n=1 | 0
  Week 78, ItoG4; n=1 | 0
  Week 84, ItoG4; n=1 | 0
  WD/study conclusion, ItoG4; n=48 | 0
  Worst-case on-therapy, ItoG4; n=65 | 1

22. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4) in Toxicity Grades for Hemoglobin at the Indicated Time Points
Description: Blood samples were collected for the evaluation of hemoglobin. Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For hemoglobin: G 1 (<LLN to 10 g/dL), mild; G 2 (<10.0 to 8.0 g/dL), moderate; G 3 (<8.0 to 6.5 g/dL), severe; G 4 (<6.5 g/dL), life threatening/disabling; G 5 (death), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 65
participants
  Week 1, AGI; n=62 | 10
  Week 2, AGI; n=64 | 16
  Week 3, AGI; n=62 | 12
  Week 6, AGI; n=47 | 10
  Week 9, AGI; n=41 | 7
  Week 12, AGI; n=30 | 6
  Week 15, AGI; n=22 | 5
  Week 18, AGI; n=17 | 2
  Week 21, AGI; n=13 | 4
  Week 24, AGI; n=11 | 3
  Week 30, AGI; n=9 | 3
  Week 36, AGI; n=5 | 0
  Week 42, AGI; n=4 | 0
  Week 48, AGI; n=3 | 0
  Week 54, AGI; n=3 | 0
  Week 60, AGI; n=2 | 0
  Week 66, AGI; n=1 | 0
  Week 72, AGI; n=1 | 0
  Week 78, AGI; n=1 | 0
  Week 84, AGI; n=1 | 0
  Withdrawal/study conclusion, AGI; n=51 | 16
  Worst-case on-therapy, AGI; n=65 | 33
  Week 1, ItoG3; n=62 | 0
  Week 2, ItoG3; n=64 | 0
  Week 3, ItoG3; n=62 | 0
  Week 6, ItoG3; n=47 | 1
  Week 9, ItoG3; n=41 | 0
  Week 12, ItoG3; n=30 | 0
  Week 15, ItoG3; n=22 | 1
  Week 18, ItoG3; n=17 | 0
  Week 21, ItoG3; n=13 | 0
  Week 24, ItoG3; n=11 | 0
  Week 30, ItoG3; n=9 | 0
  Week 36, ItoG3; n=5 | 0
  Week 42, ItoG3; n=4 | 0
  Week 48, ItoG3; n=3 | 0
  Week 54, ItoG3; n=3 | 0
  Week 60, ItoG3; n=2 | 0
  Week 66, ItoG3; n=1 | 0
  Week 72, ItoG3; n=1 | 0
  Week 78, ItoG3; n=1 | 0
  Week 84, ItoG3; n=1 | 0
  Withdrawal/study conclusion, ItoG3; n=51 | 5
  Worst-case on-therapy, ItoG3; n=65 | 9
  Week 1, ItoG4; n=62 | 0
  Week 2, ItoG4; n=64 | 0
  Week 3, ItoG4; n=62 | 0
  Week 6, ItoG4; n=47 | 0
  Week 9, ItoG4; n=41 | 0
  Week 12, ItoG4; n=30 | 1
  Week 15, ItoG4; n=22 | 0
  Week 18, ItoG4; n=17 | 0
  Week 21, ItoG4; n=13 | 0
  Week 24, ItoG4; n=11 | 0
  Week 30, ItoG4; n=9 | 0
  Week 36, ItoG4; n=5 | 0
  Week 42, ItoG4; n=4 | 0
  Week 48, ItoG4; n=3 | 0
  Week 54, ItoG4; n=3 | 0
  Week 60, ItoG4; n=2 | 0
  Week 66, ItoG4; n=1 | 0
  Week 72, ItoG4; n=1 | 0
  Week 78, ItoG4; n=1 | 0
  Week 84, ItoG4; n=1 | 0
  Withdrawal/study conclusion, ItoG4; n=51 | 0
  Worst-case on-therapy, ItoG4; n=65 | 1

23. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4) in Toxicity Grades for Lymphocytes at the Indicated Time Points
Description: Blood samples were collected for the evaluation of lymphocytes. Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For lymphocytes: G 1, mild; G 2, moderate; G 3, severe; G 4, life threatening/disabling; G 5, death related to AE; ranges were provided by local laboratories. Change from Baseline was measured as any grade increase (AGI), increase to G 3 (ItoG3), and increase to G 4 (ItoG4). Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 16
participants
  Week 1, AGI; n=14 | 0
  Week 2, AGI; n=16 | 0
  Week 3, AGI; n=16 | 0
  Week 6, AGI; n=12 | 0
  Week 9, AGI; n=11 | 0
  Week 12, AGI; n=7 | 0
  Week 15, AGI; n=6 | 0
  Week 18, AGI; n=5 | 0
  Week 21, AGI; n=4 | 2
  Week 24, AGI; n=3 | 0
  Week 30, AGI; n=2 | 0
  Week 36, AGI; n=1 | 0
  Week 42, AGI; n=0 | 0
  Week 48, AGI; n=0 | 0
  Week 54, AGI; n=0 | 0
  Week 60, AGI; n=0 | 0
  Week 66, AGI; n=0 | 0
  Week 72, AGI; n=0 | 0
  Week 78, AGI; n=0 | 0
  Week 84, AGI; n=0 | 0
  Withdrawal/study conclusion, AGI; n=10 | 1
  Worst-case on-therapy, AGI; n=16 | 3
  Week 1, ItoG3; n=14 | 0
  Week 2, ItoG3; n=16 | 0
  Week 3, ItoG3; n=16 | 0
  Week 6, ItoG3; n=12 | 0
  Week 9, ItoG3; n=11 | 0
  Week 12, ItoG3; n=7 | 0
  Week 15, ItoG3; n=6 | 0
  Week 18, ItoG3; n=5 | 0
  Week 21, ItoG3; n=4 | 0
  Week 24, ItoG3; n=3 | 0
  Week 30, ItoG3; n=2 | 0
  Week 36, ItoG3; n=1 | 0
  Week 42, ItoG3; n=0 | 0
  Week 48, ItoG3; n=0 | 0
  Week 54, ItoG3; n=0 | 0
  Week 60, ItoG3; n=0 | 0
  Week 66, ItoG3; n=0 | 0
  Week 72, ItoG3; n=0 | 0
  Week 78, ItoG3; n=0 | 0
  Week 84, ItoG3; n=0 | 0
  Withdrawal/study conclusion, ItoG3; n=10 | 0
  Worst-case on-therapy, ItoG3; n=16 | 0
  Week 1, ItoG4; n=14 | 0
  Week 2, ItoG4; n=16 | 0
  Week 3, ItoG4; n=16 | 0
  Week 6, ItoG4; n=12 | 0
  Week 9, ItoG4; n=11 | 0
  Week 12, ItoG4; n=7 | 0
  Week 15, ItoG4; n=6 | 0
  Week 18, ItoG4; n=5 | 0
  Week 21, ItoG4; n=4 | 0
  Week 24, ItoG4; n=3 | 0
  Week 30, ItoG4; n=2 | 0
  Week 36, ItoG4; n=1 | 0
  Week 42, ItoG4; n=0 | 0
  Week 48, ItoG4; n=0 | 0
  Week 54, ItoG4; n=0 | 0
  Week 60, ItoG4; n=0 | 0
  Week 66, ItoG4; n=0 | 0
  Week 72, ItoG4; n=0 | 0
  Week 78, ItoG4; n=0 | 0
  Week 84, ItoG4; n=0 | 0
  Withdrawal/study conclusion, ItoG4; n=10 | 0
  Worst-case on-therapy, ItoG4; n=16 | 0

24. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4) in Toxicity Grades for Total Neutrophils at the Indicated Time Points
Description: Blood samples were collected for the evaluation of total neutrophils. Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For neutrophils: G 1 (<LLN to 1500/millimeters cubed [mm^3] of blood plasma [bp]), mild; G 2 (<1500 to 1000/mm^3 of bp), moderate; G 3 (<1000 to 500/mm^3 of bp), severe; G 4 (<500/mm^3 of bp), life threatening/disabling; G 5 (death), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 17
participants
  Week 1, AGI; n=15 | 0
  Week 2, AGI; n=17 | 1
  Week 3, AGI; n=17 | 1
  Week 6, AGI; n=12 | 1
  Week 9, AGI; n=11 | 1
  Week 12, AGI; n=7 | 1
  Week 15, AGI; n=6 | 1
  Week 18, AGI; n=5 | 1
  Week 21, AGI; n=4 | 2
  Week 24, AGI; n=3 | 0
  Week 30, AGI; n=2 | 0
  Week 36, AGI; n=1 | 0
  Week 42, AGI; n=0 | 0
  Week 48, AGI; n=0 | 0
  Week 54, AGI; n=0 | 0
  Week 60, AGI; n=0 | 0
  Week 66, AGI; n=0 | 0
  Week 72, AGI; n=0 | 0
  Week 78, AGI; n=0 | 0
  Week 84, AGI; n=0 | 0
  Withdrawal/study conclusion,, AGI; n=12 | 1
  Worst-case on-therapy, AGI; n=17 | 3
  Week 1, ItoG3; n=15 | 0
  Week 2, ItoG3; n=17 | 0
  Week 3, ItoG3; n=17 | 0
  Week 6, ItoG3; n=12 | 0
  Week 9, ItoG3; n=11 | 0
  Week 12, ItoG3; n=7 | 0
  Week 15, ItoG3; n=6 | 0
  Week 18, ItoG3; n=5 | 0
  Week 21, ItoG3; n=4 | 0
  Week 24, ItoG3; n=3 | 0
  Week 30, ItoG3; n=2 | 0
  Week 36, ItoG3; n=1 | 0
  Week 42, ItoG3; n=0 | 0
  Week 48, ItoG3; n=0 | 0
  Week 54, ItoG3; n=0 | 0
  Week 60, ItoG3; n=0 | 0
  Week 66, ItoG3; n=0 | 0
  Week 72, ItoG3; n=0 | 0
  Week 78, ItoG3; n=0 | 0
  Week 84, ItoG3; n=0 | 0
  Withdrawal/study conclusion, ItoG3; n=12 | 0
  Worst-case on-therapy, ItoG3; n=17 | 0
  Week 1, ItoG4; n=15 | 0
  Week 2, ItoG4; n=17 | 0
  Week 3, ItoG4; n=17 | 0
  Week 6, ItoG4; n=12 | 0
  Week 9, ItoG4; n=11 | 0
  Week 12, ItoG4; n=7 | 0
  Week 15, ItoG4; n=6 | 0
  Week 18, ItoG4; n=5 | 0
  Week 21, ItoG4; n=4 | 0
  Week 24, ItoG4; n=3 | 0
  Week 30, ItoG4; n=2 | 0
  Week 36, ItoG4; n=1 | 0
  Week 42, ItoG4; n=0 | 0
  Week 48, ItoG4; n=0 | 0
  Week 54, ItoG4; n=0 | 0
  Week 60, ItoG4; n=0 | 0
  Week 66, ItoG4; n=0 | 0
  Week 72, ItoG4; n=0 | 0
  Week 78, ItoG4; n=0 | 0
  Week 84, ItoG4; n=0 | 0
  Withdrawal/study conclusion, ItoG4; n=12 | 0
  Worst-case on-therapy, ItoG4; n=17 | 0

25. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4) in Toxicity Grades for Platelet Count at the Indicated Time Points
Description: Blood samples were collected for the evaluation of platelet count. Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For platelet count: G 1 (<LLN to 75000/mm^3 of blood plasma [bp]), mild; G 2 (<75000 to 50000/mm^3 of bp), moderate; G 3 (<50000 to 25000/mm^3 of bp), severe; G 4 (<25000/mm^3 of bp), life threatening/disabling; G 5 (death), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 65
participants
  Week 1, AGI; n=62 | 1
  Week 2, AGI; n=64 | 2
  Week 3, AGI; n=62 | 0
  Week 6, AGI; n=47 | 2
  Week 9, AGI; n=41 | 3
  Week 12, AGI; n=30 | 2
  Week 15, AGI; n=22 | 2
  Week 18, AGI; n=17 | 0
  Week 21, AGI; n=13 | 1
  Week 24, AGI; n=11 | 0
  Week 30, AGI; n=9 | 2
  Week 36, AGI; n=5 | 0
  Week 42, AGI; n=4 | 0
  Week 48, AGI; n=3 | 0
  Week 54, AGI; n=3 | 0
  Week 60, AGI; n=2 | 0
  Week 66, AGI; n=1 | 0
  Week 72, AGI; n=1 | 0
  Week 78, AGI; n=1 | 0
  Week 84, AGI; n=1 | 0
  Withdrawal/study conclusion, AGI; n=51 | 4
  Worst-case on-therapy, AGI; n=65 | 10
  Week 1, ItoG3; n=62 | 0
  Week 2, ItoG3; n=64 | 0
  Week 3, ItoG3; n=62 | 0
  Week 6, ItoG3; n=47 | 0
  Week 9, ItoG3; n=41 | 0
  Week 12, ItoG3; n=30 | 0
  Week 15, ItoG3; n=22 | 0
  Week 18, ItoG3; n=17 | 0
  Week 21, ItoG3; n=13 | 0
  Week 24, ItoG3; n=11 | 0
  Week 30, ItoG3; n=9 | 0
  Week 36, ItoG3; n=5 | 0
  Week 42, ItoG3; n=4 | 0
  Week 48, ItoG3; n=3 | 0
  Week 54, ItoG3; n=3 | 0
  Week 60, ItoG3; n=2 | 0
  Week 66, ItoG3; n=1 | 0
  Week 72, ItoG3; n=1 | 0
  Week 78, ItoG3; n=1 | 0
  Week 84, ItoG3; n=1 | 0
  Withdrawal/study conclusion, ItoG3; n=51 | 0
  Worst-case on-therapy, ItoG3; n=65 | 1
  Week 1, ItoG4; n=62 | 0
  Week 2, ItoG4; n=64 | 0
  Week 3, ItoG4; n=62 | 0
  Week 6, ItoG4; n=47 | 0
  Week 9, ItoG4; n=41 | 0
  Week 12, ItoG4; n=30 | 0
  Week 15, ItoG4; n=22 | 0
  Week 18, ItoG4; n=17 | 0
  Week 21, ItoG4; n=13 | 0
  Week 24, ItoG4; n=11 | 0
  Week 30, ItoG4; n=9 | 0
  Week 36, ItoG4; n=5 | 0
  Week 42, ItoG4; n=4 | 0
  Week 48, ItoG4; n=3 | 0
  Week 54, ItoG4; n=3 | 0
  Week 60, ItoG4; n=2 | 0
  Week 66, ItoG4; n=1 | 0
  Week 72, ItoG4; n=1 | 0
  Week 78, ItoG4; n=1 | 0
  Week 84, ItoG4; n=1 | 0
  Withdrawal/study conclusion, ItoG4; n=51 | 0
  Worst-case on-therapy, ItoG4; n=65 | 0

26. Secondary Outcome: Number of Participants With Change From Baseline (Measured as AGI, ItoG3, and ItoG4) in Toxicity Grades for White Blood Cell (WBC) Count at the Indicated Time Points
Description: Blood samples were collected for the evaluation of WBC count. Toxicity was measured in grades (AE severity) per NCI CTCAE, v3.0, displaying Grades (G) 1-5 with unique clinical descriptions of the severity of each AE. For WBCs: G 1 (<LLN to 3000/mm^3 of blood plasma [bp]), mild; G 2 (<3000 to 2000/mm^3 of bp), moderate; G 3 (<2000 to 1000/mm^3 of bp), severe; G 4 (<1000/mm^3 of bp), life threatening/disabling; G 5 (death), death related to AE. Worst-case on-therapy reflects the most severe change at any time point measured post treatment.
Time Frame: as for outcome 11
Population: Safety Population. Only those participants with data available at the specified time points were evaluated.
Measure: Number; unit: participants
Arm/Group | Lapatinib + Capecitabine
Number analyzed (Participants) | 65
participants
  Week 1, AGI; n=62 | 5
  Week 2, AGI; n=64 | 9
  Week 3, AGI; n=62 | 6
  Week 6, AGI; n=47 | 5
  Week 9, AGI; n=41 | 3
  Week 12, AGI; n=30 | 7
  Week 15, AGI; n=22 | 4
  Week 18, AGI; n=17 | 3
  Week 21, AGI; n=13 | 3
  Week 24, AGI; n=11 | 1
  Week 30, AGI; n=9 | 3
  Week 36, AGI; n=5 | 2
  Week 42, AGI; n=4 | 2
  Week 48, AGI; n=3 | 1
  Week 54, AGI; n=3 | 1
  Week 60, AGI; n=2 | 0
  Week 66, AGI; n=1 | 0
  Week 72, AGI; n=1 | 0
  Week 78, AGI; n=1 | 0
  Week 84, AGI; n=1 | 0
  Withdrawal/study conclusion, AGI; n=51 | 2
  Worst-case on-therapy, AGI; n=65 | 17
  Week 1, ItoG3; n=62 | 0
  Week 2, ItoG3; n=64 | 0
  Week 3, ItoG3; n=62 | 0
  Week 6, ItoG3; n=47 | 0
  Week 9, ItoG3; n=41 | 0
  Week 12, ItoG3; n=30 | 1
  Week 15, ItoG3; n=22 | 0
  Week 18, ItoG3; n=17 | 0
  Week 21, ItoG3; n=13 | 0
  Week 24, ItoG3; n=11 | 0
  Week 30, ItoG3; n=9 | 0
  Week 36, ItoG3; n=5 | 0
  Week 42, ItoG3; n=4 | 0
  Week 48, ItoG3; n=3 | 0
  Week 54, ItoG3; n=3 | 0
  Week 60, ItoG3; n=2 | 0
  Week 66, ItoG3; n=1 | 0
  Week 72, ItoG3; n=1 | 0
  Week 78, ItoG3; n=1 | 0
  Week 84, ItoG3; n=1 | 0
  Withdrawal/study conclusion, ItoG3; n=51 | 0
  Worst-case on-therapy, ItoG3; n=65 | 1
  Week 1, ItoG4; n=62 | 0
  Week 2, ItoG4; n=64 | 0
  Week 3, ItoG4; n=62 | 0
  Week 6, ItoG4; n=47 | 0
  Week 9, ItoG4; n=41 | 0
  Week 12, ItoG4; n=30 | 0
  Week 15, ItoG4; n=22 | 0
  Week 18, ItoG4; n=17 | 0
  Week 21, ItoG4; n=13 | 0
  Week 24, ItoG4; n=11 | 0
  Week 30, ItoG4; n=9 | 0
  Week 36, ItoG4; n=5 | 0
  Week 42, ItoG4; n=4 | 0
  Week 48, ItoG4; n=3 | 0
  Week 54, ItoG4; n=3 | 0
  Week 60, ItoG4; n=2 | 0
  Week 66, ItoG4; n=1 | 0
  Week 72, ItoG4; n=1 | 0
  Week 78, ItoG4; n=1 | 0
  Week 84, ItoG4; n=1 | 0
  Withdrawal/study conclusion, ItoG4; n=51 | 0
  Worst-case on-therapy, ItoG4; n=65 | 0

ADVERSE EVENTS:
Arm/Group | Lapatinib + Capecitabine
Serious Adverse Events (participants affected / at risk) | 22/67
Other Adverse Events (participants affected / at risk) | 63/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib + Capecitabine (N=67)
Vomiting (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Poisoning (Injury, poisoning and procedural complications) | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 1
Embolism (Vascular disorders) | 1
Ejection fraction decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib + Capecitabine (N=67)
Diarrhea (Gastrointestinal disorders) | 27
Decreased appetite (Metabolism and nutrition disorders) | 23
Fatigue (General disorders) | 23
Nausea (Gastrointestinal disorders) | 23
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 17
Anemia (Blood and lymphatic system disorders) | 16
Abdominal pain (Gastrointestinal disorders) | 13
Abdominal pain upper (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 11
Weight decreased (Investigations) | 11
Rash (Skin and subcutaneous tissue disorders) | 10
Aspartate aminotransferase increased (Investigations) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dizziness (Nervous system disorders) | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Alanine aminotransferase increased (Investigations) | 8
Constipation (Gastrointestinal disorders) | 8
Edema peripheral (General disorders) | 8
Stomatitis (Gastrointestinal disorders) | 8
Pyrexia (Gastrointestinal disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Insomnia (Psychiatric disorders) | 6
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 6
Blood creatinine increased (Investigations) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 5
Pain (General disorders) | 5
Abdominal discomfort (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Hemoglobin decreased (Blood and lymphatic system disorders) | 4
Headache (Nervous system disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 4
Mouth ulceration (Gastrointestinal disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.